CLINICAL TRIAL: NCT06773975
Title: A 12-week Pilot Randomized Controlled Trial of an Oral Nutritional Supplement in Improving the Nutritional and Health Outcomes of the Elderly in Peri Urban Communities of the La Nkwantanang Madina Municipality in the Greater Accra Region
Brief Title: The Effect of an Oral Nutritional Supplement on the Nutritional and Health Outcomes of the Elderly
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Ghana (Other)
Responsible Party: Principal Investigator, Matilda Anim-Fofie, Principal Investigator and a PhD candidate studying Nutrition at the Department of Nutrition and Food Science-University of Ghana, University of Ghana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ORTONSINTUGDNFSSFPEMATGLSTJOSA
Record Dates: First submitted 2024-11-21; First posted 2025-01-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Hand Grip Strength; Body Weight; Iron Deficiency; Anaemia; Total Cholesterol; Protein Deficiency
Keywords: Nutritional and health outcomes; Oral Nutritional Supplement; Elderly; Peri urban; Randomized Controlled Trial
MeSH Terms: conditions — Hypertension; Body Weight; Iron Deficiencies; Anemia; Protein Deficiency | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: The study participants will be randomized to two arms; one arm will be given a plant-based oral nutritional supplement for 12 weeks and the other arm (control) will not be given any treatment.
  An oral nutritional supplement arm and a no treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral nutritional supplement (Experimental): Participants will consume daily for 12 weeks in between meals, a 300 ml oral nutritional supplement
  Interventions: Dietary Supplement: Oral nutritional supplementation
- No treatment or the control group (No Intervention): The participants in the no treatment group or control group will not receive any treatment during the 12 weeks except for nutrition education that will be given at certain points to all the participants

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplementation — The oral nutritional supplement is a locally made plant based formulation targeted to improve the nutritional status of the elderly
  Arms: Oral nutritional supplement

SUMMARY:
I am conducting this research to find out if a peanut based food that is ready to use would improve the nutritional and health outcomes of the elderly when they consume it daily for 12 weeks. Eligible participants will be assigned randomly to any of these 2 groups.

1. To consume the food once a day in between meals in addition to their usual food for 12 weeks (3 months) or
2. A control group that will not be given the food. Measurements such as weight, blood pressure and the hand grip strength will be taken at the certain points of the study. A sterile needle will be used to draw about 5 ml of venous blood (from the arm) at the beginning of the study and after 12 weeks. Analyses would be carried out on the blood to know if the food has made an impact on serum albumin, ferritin, haemoglobin and cholesterol. If the findings of the study are favourable, it would provide insights for a larger randomized controlled trial that could establish the efficacy of a locally produced peanut based food for the feeding of the elderly.

DETAILED DESCRIPTION:
Study design A hybrid study comprising of a cross sequential study and a randomized controlled trial.

Study area The study locations are the following five peri urban communities out of the ten peri urban communities in the La Nkwantanang Madina Municipality (LANMA) of the Greater Accra Region in Ghana; Ayi Mensah, Kweiman, Danfa, Adoteiman and Otinibi. These have been conveniently selected because they are a continuous stretch of five communities in the order listed above to reduce the cost of transportation of data collectors and logistics, distribution of the intervention and data collection based on funds available for the project.

Sample size Assumptions: A Cohen's medium effect size of 0.3, a statistical power of 80% at a 5% level of significance, G-power 3.9.1.7 software generated a sample size of 90 participants per treatment group. Accounting for attrition rate + loss to follow up of 10% = 99 participants * 2 treatment groups

= A total sample size of 198 elderly individuals. This has been rounded off to 200 participants. The census to recruit the 200 eligible participants has been completed as of December 13, 2024.

A cross-sectional survey to identify the relationship between usual dietary intake, handgrip strength and blood pressure has been conducted for the 200 participants. Eighty of the participants will be randomly selected as participants for a 12 week randomized control trial.

Assumptions (80 participants): A Cohen's medium effect size of 0.25, a statistical power of 90% at a 5% level of significance, GPower 3.1.9.4 generated a sample size of 36 participants per treatment group. Accounting for attrition rate and a loss to follow up of 10% = 40 participants * 2 treatment groups. A total sample size of 80 elderly individuals.

Data collection for the randomized control trial An interviewer administered questionnaire will be used to obtain the following information at different points of assessments

Baseline data collection Sociodemographic characteristics and medical history such as age, sex, highest level of education, marital status, ethnicity and use of iron supplements, anti-hypertensive drugs and cholesterol lowering drugs will be collected.

Baseline, midline (6 weeks) and endline (12 weeks) A multiple pass quantitative 24-hour dietary recall to obtain information on dietary intake. Household measures and food models will be used to estimate portion sizes. The Physical Activity Scale for the Elderly (PASE) by Washburn et al. (1993) will be used to measure level of physical activity. Body weight, hand grip strength, systolic and diastolic blood pressure will be measured.

Weekly All participants will receive nutrition education at baseline and weekly thereafter. Information on adherence will be collected by evidence of pouches of previous week's ration to calculate percentage of quantity consumed. The 24-hour dietary recall will also be used to track adherence. Information on morbidity on the use of oral nutritional supplements will be collected using the questionnaire for gastrointestinal problems adapted from Pereira et al. (2014).

Baseline and 12 weeks A qualified phlebotomist will take a 5ml venous blood for analyses of the following: serum albumin, serum ferritin, serum cholesterol and haemoglobin

The intervention A 7-day ration of the oral nutritional supplement will be distributed to the intervention arm once a week. A day's serving of 330 ml is to be consumed in between meals. After endline data collection, the control arm will be given a ration of the oral nutritional supplement that will be enough for one month.

Statistical analyses

* To investigate the effect of sociodemographic characteristics, dietary intake and level of physical activity on the outcome measures, binary logistic regression for categorical variables, multinomial or ordinal logistics regression for multiple variables and linear regression for continuous variables
* To determine the efficacy of the oral nutritional supplement on outcome measures within the same treatment arm, repeated measures ANOVA and paired-sample t-test will be used
* To determine the differences in outcomes between the treatment groups the multivariate ANOVA and independent sample t-test will be used.

Data entry and management Field investigators will enter data collected on pre-programmed tablets that are functioning well. After each day's work, the supervisor will cross check and review all data in the presence of field investigators to ensure that complete and consistent data is finally submitted. The supervisor will flag any aberrant values and consult with the relevant field worker within 24 hours so that gaps will be filled, errors resolved and repeat interviews/visits can be conducted if need be. The submitted data will be accessed by the principal investigator daily for real-time review and monitoring. Once all data have been entered, reviewed and cleaned, final SPSS datasets will be generated and made available to the principal investigator for analysis. As soon as the manuscripts summarizing the study's primary outcomes are published, all datasets will be made available to any one who request it for research purposes.

Informed consent forms will be stored under lock and key.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals aged 60 years and above
* Consent to participate

Exclusion Criteria:

* Peanut allergy
* Millet allergy
* Sesame seeds allergy
* The use of oral nutritional supplement
* Sickle cell disease
* End stage and terminal illness (cancer, stroke, liver disease, dialysis)
* Clinical depression
* Speech impairment
* Hearing impairment
* Visual impairment
* Cognitive impairment Screening/for cognitive impairment; the Abbreviated Mental Test Score by HODKINSON (1972) was adapted for use.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum albumin in g/dL; a change in the concentration of serum albumin from baseline to 12 weeks | Measurement will be taken at baseline (before commencement of intervention) and after 12 weeks of intervention
  A phlebotomist will draw 5 ml of venous blood in the morning after a 12 hour overnight fast from each participant for analysis in the laboratory. This will be done at baseline and after 12 weeks. Generally the reference values for serum albumin level is 3.5 g/dL to 5.5 g/dL, however there could be slight differences for the range depending on the laboratory. Analyses will be carried out to ascertain any change in serum albumin levels between baseline and at 12 weeks. Comparisons will be made to ascertain the differences between the serum albumin concentration of the experimental arm and the no intervention arm at baseline and at 12 weeks. Participants with a serum albumin concentration below the reference range will be classified as having low serum albumin concentration.
Body weight measured in kilograms to determine the change in weight at 3 different points of measurements within the 12 weeks of commencement of intervention | At baseline, midline (6 weeks) and endline (12 weeks)
  The participants will be weighed in light clothing and without shoes. They will be instructed to stand up straight as possible, with heels close together, legs straight as possible, arms at the sides and shoulders relaxed. Body weight will be recorded to the nearest 0.1 kg. Two weight readings will be taken, however a third reading will be taken if the first two readings differ by more than 0.1kilogram. Periodically, the scale will be calibrated for accuracy. Body weight of each participant will be measured at baseline (before the commencement of the intervention), 6 weeks and 12 weeks. Analyses will be done to find out the trend in change in the body weight along the 3 different points of measurement. Comparisons will be made between the experimental group and the no intervention group at each point of measurement

SECONDARY OUTCOMES:
Haemoglobin level in g/dl to determine the prevalence of anaemia at baseline and after 12 weeks | Haemoglobin level measured at baseline (before the intervention) and after 12 weeks
  A phlebotomist will draw 5 ml of venous blood in the morning after a 12 hour overnight fast from each participant for analysis in the laboratory to measure the concentration of haemoglobin in mg/dL at baseline and after 12 weeks. The World Health Organization reference values for anaemia in elderly men is haemoglobin level below 13g/dL and for elderly women, haemoglobin level below 12g/dL. Analyses will be carried out to ascertain the prevalence of anaemia at baseline and 12 weeks. Comparisons will be made to determine the differences in the prevalence of anaemia between the experimental arm and the no intervention arm.
Concentration of serum ferritin in µg/l to determine the prevalence of iron deficiency at baseline and at 12 weeks | Baseline and after 12 weeks
  A phlebotomist will draw 5 ml of venous blood in the morning after a 12 hour overnight fast from each participant for analysis in the laboratory to measure the concentration of serum ferritin in µg/L at baseline and at 12 weeks. The WHO reference values for iron deficiency in apparently healthy elderly persons (60 years and above) is serum ferritin concentration less than 5 µg/L and for those with infections and inflammation, less than 70µg/L . Analyses will be carried out to ascertain the prevalence of iron deficiency at baseline and 12 weeks. Comparisons will be made to know the differences in the prevalence of iron deficiency between the experimental arm and the no intervention arm at baseline and after 12 weeks
Total serum cholesterol measured in mg/dL at baseline and at 12 weeks to determine the change in total serum cholesterol | Baseline and after 12 weeks
  A phlebotomist will draw 5 ml of venous blood after a 12 hour overnight fast to measure the concentration of total serum cholesterol in mg/dl for all participants at baseline before the intervention and after 12 weeks. Generally, a normal total serum cholesterol level for adults is < 200 mg/dL, borderline high is 200 to 239 mg/dL and high is 240 mg/dL and above. Analyses will be done to know the percentage of participants who have normal, borderline high and high total serum cholesterol at baseline and at endline at 12 weeks. Comparison will be made between the experimental arm and the intervention arm to ascertain the differences in the change in their total serum cholesterol
Hand grip strength of the dominant arm measured in kilograms to determine the change in handgrip strength at 3 different points of measurements; At baseline, midline (6 weeks) and endline (12 weeks) | At baseline, midline (6 weeks) and endline (12 weeks)
  Each participant will sit on chair and with the dynamometer in the hand, position his or her dominant arm at the elbow bent at a 90-degree angle and squeeze the dynamometer as hard as possible for 3 seconds and apply a grip force in a smooth motion to avoid jerking. The reading will be taken in kilograms. This will be repeated twice more for a total of three readings. The average of the three readings is the hand grip strength. Analyses will be done to find out the trend in change in the handgrip strength along the 3 different points of measurement (baseline, 6 weeks and at 12 weeks). Comparisons will be made between the experimental group and the no intervention group at each point of measurement.
Systolic and diastolic blood pressure measured in mmHg to determine the prevalence of elevated blood pressure at baseline, midline (6 weeks) and endline (12 weeks) | At baseline, midline (6 weeks) and endline (12 weeks)
  Participants will sit in a rested position and blood pressure will be measured after a 5 minute rest using a digital sphygmomanometer. The mean of two readings to the nearest mmHg will be recorded. A third reading will be taken if the difference in the first two readings is more than 10mmHg. There will be a 2 minute rest in between measurements. The approved definition of high blood pressure by the WHO is a level of systolic blood pressure of 140 mmHg or more or a level of diastolic blood pressure of 90 mmHg or more. Analyses will be done to find out the trend in change in the blood pressure along the 3 different points of measurement (baseline, 6 weeks and at 12 weeks). Comparisons will be made between the experimental group and the no intervention group at each point of measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria E. Otoo, PhD in Nutrition, Study Director — University of Ghana; Matilda Steiner-Asiedu, PhD in Nutrition, Study Director — University of Ghana; Jolene Nyako, PhD in Nutrition, Study Director — Council for Scientific and Industrial Research-Food Research Institute, Accra-Ghana; Firibu K. Saalia, PhD in Food Science, Study Director — University of Ghana
Locations (1):
- University of Ghana, Accra, Greater Accra Region, Ghana

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD and all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: As soon as the manuscripts summarizing the study's outcomes are published, all datasets will be made available to any one who request it for research purposes (beginning 6 months after publication) with no end date
Access Criteria: All publications will bear the email address of the principal investigator/corresponding author of the publication. Anyone who would want to obtain the IPD could contact the corresponding author or the principal investigator. The one making the request would submit a proposal of what he intends to use the data for and the type of analyses that would be done. All correspondence and submissions will be via email.
  Requests for sharing of IPD will be reviewed by the sponsors and collaborators of this study.

REFERENCES:
- [Background] Billingham et al. 2013
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031